CLINICAL TRIAL: NCT07255521
Title: Effects of a Prehabilitation Program on Frailty, Function, Quality of Life, and Post-Transplant Outcomes in Candidates for Hematopoietic Stem Cell Transplantation: A Randomized Clinical Trial
Brief Title: Prehabilitation to Improve Frailty, Function, and Quality of Life in Candidates for Hematopoietic Stem Cell Transplantation
Acronym: PREHAB-HSCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Salvador (Other)
Collaborators: Universidad Católica del Maule (Other); University of Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: hsalvador
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: Prehabilitation; Hematologic Malignancies; Frailty; Cancer-Related Frailty; Functional capacity; Physical Function; Quality of life; Post-Transplant Outcomes
MeSH Terms: conditions — Hematologic Neoplasms; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor is masked to group allocation. Participants, care providers, and investigators are not masked due to the nature of the behavioral intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation Program (Experimental): Participants in this arm will receive a multimodal prehabilitation program that includes supervised aerobic and resistance exercise, balance and flexibility training, respiratory exercises, education on healthy lifestyle behaviors, and occupational therapy. The intervention is delivered in a hybrid format (in-person and remote), 2-3 sessions per week for 15-18 sessions in total.
  Interventions: Other: Multimodal Prehabilitation
- Usual Care (No Intervention): Participants in this arm will receive standard medical care as determined by their clinical team. No structured prehabilitation or additional exercise-based intervention will be provided.

INTERVENTIONS:
Other: Multimodal Prehabilitation — In-Person Sessions:
  Supervised by a cancer-specialized physiotherapist. Includes:
  * Aerobic exercise: 20-25 min. at moderate intensity (BORG 4-6 or 60-80% HRmax).
  * Resistance training: 20-25 min. at 10-12 RM, using dumbbells or resistance bands.
  * Flexibility or balance training: 5 minutes.
  * Warm-up and cool-down: 5 minutes each.
  Sessions last 1-1.5 hours, 2-3 times/week, 15-18 sessions Education on healthy habits, smoking and alcohol cessation, sleep hygiene, and physical activity.
  Daily home-exercise logs and telephone supervision will support adherence.
  Remote Sessions:
  (Video call/Zoom, 45-60 min): Mixed exercises, breathing techniques, and incentive spirometry.
  Occupational Therapy Intervention
  * cognitive training (memory, attention, executive function),
  * upper limb functional training (fine/gross motor skills, bilateral coordination, prehension)
  * ADL/IADL training
  * energy-conservation techniques and joint-protection strategies. 6-8 sessions, 30-45 min.
  Other Names: Exercise Intervention; Occupational Therapy Intervention
  Arms: Prehabilitation Program

SUMMARY:
Candidates for hematopoietic stem cell transplantation (HSCT) frequently experience declines in strength, physical function, and quality of life before the procedure. Many also present fatigue, limitations in daily activities, and an increased risk of complications during and after hospitalization. Optimizing physical condition before transplantation may improve post-procedure recovery.

This study will evaluate whether a prehabilitation program improves physical function, frailty, and quality of life in adults preparing for HSCT. The intervention consists of supervised exercise, education, and activities designed to enhance endurance and functional capacity. Although prehabilitation has shown benefits in other oncologic populations, it has been minimally studied in HSCT candidates, and no structured programs have been evaluated in Chile.

A total of 68 adults will be randomly assigned to a prehabilitation group or a usual-care control group. The prehabilitation group will receive a personalized program including aerobic and resistance exercise, stretching, balance training, respiratory exercises, and education on healthy behaviors, delivered through a hybrid model of in-person and remote sessions. Occupational therapy will also be provided to support functional and cognitive abilities. The control group will continue with standard medical care.

Baseline and post-intervention assessments will include measures of strength, frailty, fatigue, balance, cognitive function, daily activities, and quality of life. Post-transplant outcomes such as hospital length of stay, complications, and readmissions within three months will also be recorded. Feasibility, adherence, satisfaction, and adverse events will be evaluated.

Findings from this trial may inform the development of structured prehabilitation programs for HSCT candidates and support the implementation of evidence-based supportive care strategies in hematologic oncology.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is a complex treatment widely used for hematologic malignancies. Although it offers curative potential, many patients experience significant declines in physical functioning, increased frailty, fatigue, and reduced quality of life before and after transplantation. Lower functional reserve prior to HSCT has been associated with greater treatment-related complications, longer hospital stays, and slower recovery. Despite growing evidence supporting exercise-based interventions in cancer care, prehabilitation has been minimally studied in HSCT candidates, and no structured prehabilitation program has been tested in Chile.

This randomized clinical trial investigates whether a multimodal prehabilitation program delivered before HSCT can improve frailty, functional capacity, quality of life, and early post-transplant outcomes. The intervention combines supervised aerobic and resistance exercise, balance and flexibility training, respiratory exercises, education on healthy behaviors, and a structured home-based component. A hybrid delivery model (in-person and remote sessions) allows tailoring to individual needs and supports continuity of care. Occupational therapy sessions complement the program by addressing cognitive and functional abilities relevant to daily activities.

A total of 68 adults preparing for HSCT will be randomized in a 1:1 ratio to either the prehabilitation group or a usual-care control group. The study uses concealed allocation and blinded outcome assessment. Feasibility-including adherence, acceptability, and reported adverse events-will also be evaluated to determine whether the program can be safely and efficiently implemented in a real-world transplant setting.

The results of this trial will provide new evidence on whether prehabilitation can strengthen physical resilience before HSCT, reduce early post-transplant complications, and support better recovery. Findings may guide the development of standardized prehabilitation programs for patients undergoing HSCT and inform national recommendations for supportive care in hematologic oncology.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Diagnosis of hematologic malignancy requiring HSCT (autologous or allogeneic).
* Minimum of ≥4 weeks available before the scheduled transplant.
* "Pre-frail" or "frail" according to the HCT Frailty Scale.
* ECOG ≤2 or Karnofsky ≥60.
* Internet access (videocalls, Zoom platform, or a facilitator) for remote sessions.

Exclusion Criteria:

* Cognitive impairment preventing questionnaire completion.
* Musculoskeletal comorbidities preventing participation in supervised exercise-based prehabilitation.
* Prior chemotherapy or radiotherapy not related to the hematologic malignancy.
* Medical conditions limiting participation (e.g., unstable angina, arrhythmia, hypertension or heart failure, acute systemic infection with fever, acute myocarditis, or pericarditis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-12-26 (Estimated); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | Baseline and post-intervention (4-6 weeks)
  In the 1-minute Sit-to-Stand Test (1-min STST), participants perform repeated sit-to-stand movements for 60 seconds. The number of repetitions completed will be record. Higher scores indicate better functional capacity. The test is validated as a measure of submaximal functional endurance.
Frailty | Baseline and immediately post-intervention (approximately 4-6 weeks).
  Frailty will be assessed using the Hematopoietic Cell Transplantation-Comorbidity Index Frailty Scale (HCT Frailty Scale). The scale includes 8 items: Clinical Frailty Scale (CFS), Instrumental Activities of Daily Living (IADL), Self-Rated Health Question, Falls history, Handgrip strength, Timed Up and Go Test (TUG), serum albumin levels, and C-reactive protein (CRP). Each item is scored as normal or abnormal, yielding a total score from 0 to 10.5, with higher scores indicating greater frailty. Participants will be classified as fit, pre-frail, or frail.
Lower Limb Strength | Baseline and post-intervention (4-6 weeks)
  In the 30-second Sit-to-Stand Test (30s STST), participants are instructed to stand up and sit down from a standard chair as many times as possible within 30 seconds. The total number of completed repetitions is recorded, with higher numbers indicating better lower-limb strength. The test has demonstrated good reliability in cancer and older adult populations.
Handgrip Strength | Baseline and post-intervention (4-6 weeks)
  Handgrip strength will be assessed with the Jamar® hydraulic hand dynamometer following the American Society of Hand Therapists standardized protocol. The maximum isometric grip force (in kilograms) will be recorded. Reduced grip strength is associated with frailty and poor outcomes in cancer populations.
Fatigue | Baseline and post-intervention (4-6 weeks)
  Fatigue will be assessed using the Brief Fatigue Inventory (BFI), a validated 9-item questionnaire evaluating fatigue severity and functional interference on a 0-10 numeric scale. The instrument provides a global fatigue score, categorized as: 0 (no fatigue), 1-3 (mild), 4-6 (moderate), and 7-10 (severe). Higher scores indicate greater fatigue.
Dynamic Balance and Fall Risk | Baseline and post-intervention (4-6 weeks)
  Dynamic balance and fall risk will be assessed using the Timed Up and Go Test (TUG). Participants stand up from a chair, walk 3 meters, turn, return, and sit down. The time (in seconds) to complete the task is recorded. Faster times indicate better mobility and lower fall risk. A time ≤10 seconds is considered normal functional mobility.
Subjective physical activity level | Baseline and post-intervention (4-6 weeks)
  Physical activity levels will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). The instrument records walking, moderate-intensity, and vigorous-intensity activities performed during the previous 7 days. Data are converted into metabolic equivalent minutes per week (MET-min/week). Higher scores represent higher physical activity levels.
Objective Physical Activity | 7-day monitoring at baseline and 7-day monitoring post-intervention
  It will be measured using an ActivPAL™ accelerometer, recording steps, cadence, posture, transitions, moderate-intensity activity, and sedentary behavior over 10 days.
Post-Transplant Outcomes | During index hospitalization for HSCT
  It includes:
  * Hospital length of stay: days from stem cell infusion to discharge.
  * Post-transplant complications (within 3 months).
  * Hospital readmission: number and duration of readmissions within 3 months.

SECONDARY OUTCOMES:
Cognitive Function | Baseline and post-intervention (4-6 weeks)
  Cognitive function will be evaluated using the Mini-Mental Abbreviated Test validated for Chile. The instrument assesses orientation, memory, attention, calculation, and language, with a maximum score of 35. Scores ≥30 indicate normal cognition; lower scores reflect mild to severe cognitive impairment.
Functioning and Disability | Baseline and post-intervention (4-6 weeks)
  Disability will be assessed using the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0), a validated 36-item instrument aligned with the ICF domains. It evaluates cognition, mobility, self-care, getting along, life activities, and participation. Scores are standardized on a 0-100 scale, with higher scores indicating greater disability.
Quality of Life measured by the FACT-BMT | Baseline and post-intervention (4-6 weeks)
  Health-related quality of life will be assessed using the Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT). The questionnaire includes Physical, Social/Family, Emotional, Functional Well-Being, and Bone Marrow Transplant-Specific Concerns. Total scores range from 0 to 148, with higher scores indicating better quality of life.
Feasibility: adherence, satisfaction, and adverse events | Throughout the intervention period (4-6 weeks)
  Feasibility will be assessed through: (1) adherence (percentage of prescribed sessions completed), (2) user satisfaction measured via a 9-item Likert-scale questionnaire, and (3) number and severity of adverse events reported during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Luz Alejandra Lorca, Master, Principal Investigator — Hospital del Salvador
Locations (1):
- Hospital del Salvador, Santiago, Providencia, Chile

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because the study did not include a data-sharing plan in the protocol, and ethical approval and consent documents restrict data use to the research team only.